CLINICAL TRIAL: NCT00558090
Title: Randomised Clinical Trial of the Optimization of Procedural Pain Control in ICU Patients
Brief Title: The Optimization of Procedural Pain Control in Intensive Care Unit (ICU) Patients
Acronym: OPCIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Dr. C.A.J. Knibbe, hospital pharmacist- clinical pharmacologist, St Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-07.15A/OPCIC; NL18828.100.07
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2008-10

CONDITIONS: Critical Illness
Keywords: pain; Intensive Care Unit; morphine; pKpD; numerical rating scale; critically ill patients
MeSH Terms: conditions — Critical Illness; Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): patients receive 2,5 mg morphine iv, before the first intervention on the day after admission in the ICU
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: morphine — patients receive 7,5 mg morphine iv 30 minutes before intervention (turning of the patient), the day after admission in the ICU. before, during and after, the patient will be asked to rate the pain using the NRS

SUMMARY:
The purpose of this study is to determine the influence of morphine 2,5 mg or morphine 7,5 mg iv during a painful and unavoidable intervention in critically ill patients.

DETAILED DESCRIPTION:
In 2006, in the Intensive Care Unit (ICU) of the St. Antonius Hospital an analgesia improvement program has been implemented. This program consisted of training of ICU nurses and intensivists using a hospital based standardized pain protocol, and systematic pain measurements in rest, rated by the patient himself whenever possible or otherwise by the attending nurse. This program has resulted in a reduction of severe pain levels (NRS≥4) in ICU patients in rest from 41% to 22%. In order to further reduce this percentage, a pain titration protocol is introduced in 2007. As no attention has yet been paid to intervention-related pain levels in these patients, in this prospective study pain control will be studied using different analgesic dosages of morphine iv (2,5 mg vs 7,5 mg) around unavoidable painful interventions within a pain titration protocol for pain control in rest.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU of the St. Antonius hospital, between 18-85 years old en weighing between 45-140 kg.

Exclusion Criteria:

* Pregnancy/ breastfeeding
* Language barrier
* Known morphine iv allergy
* Comatose patients (cooled)
* Patients who are suspected to be brain-dead
* Unintubated patients on the verge of intubation due to respiratory insufficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with a NRS of ≥ 4 during intervention (2.5 mg versus 7.5 mg morphine iv) | The first intervention one day after admission

SECONDARY OUTCOMES:
The mean NRS during an intervention (2.5 mg versus 7.5 mg morphine iv) | 10 days
The percentage of patients with at least one NRS-score of ≥ 4 at rest during ICU stay | 10 days
The mean NRS per patient in rest during ICU stay | 10 days
The percentage of patients with a NRS of ≥ 6 during intervention (2.5 mg versus 7.5 mg morphine iv) | one day after admission in the ICU
Pharmacokinetic parameters of morphine iv (volumes of distribution and clearance values) | 10 days
Pharmacodynamic parameters of morphine iv (EC50 etc) | 10 days
Covariates for the PK/PD of morphine iv | 10 days
Safety and other measures of the analgesics (morphine iv and paracetamol) used for intervention related pain as well as pain titration protocol for pain control in rest. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Catherijne AJ Knibbe, Pharm D, Principal Investigator — St Antonius Hospital, Department of Clinical Pharmacy
Locations (1):
- St antonius Hospital, Nieuwegein, Netherlands

REFERENCES:
- [Derived] Goulooze SC, Krekels EH, Saleh MA, Ahlers SJ, Valitalo PA, van Dongen EP, van Schaik RH, Hankemeier T, Tibboel D, Knibbe CAJ. Predicting Unacceptable Pain in Cardiac Surgery Patients Receiving Morphine Maintenance and Rescue Doses: A Model-Based Pharmacokinetic-Pharmacodynamic Analysis. Anesth Analg. 2021 Mar 1;132(3):726-734. doi: 10.1213/ANE.0000000000005228. PMID 33122543